CLINICAL TRIAL: NCT00227110
Title: Role of Pioglitazone in the Treatment of Non-alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Kenneth Cusi, M.D., The University of Texas Health Science Center at San Antonio and the San Antonio VAMC.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTHSCSA IRB# 001-5014-331
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH, IGT, T2DM
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone 30 mg/d will be given for 8 weeks and titrated to 45 mg/d until the end of the 6-month study in a randomized, double-blind, study design.
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo once daily is given following a randomized, double-blind, placebo-controlled study design.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 30 mg/d for 8 weeks and titrated to 45 mg/d until completing 6 months of treatment.
  Other Names: Actos (Takeda Pharmaceuticals).
  Arms: Pioglitazone
Drug: Placebo — Placebo is given to match pioglitazone.
  Arms: Placebo

SUMMARY:
To determine the role of pioglitazone in the treatment of nonalcoholic steatohepatitis (NASH) in patients with glucose intolerance or type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
v. 4/1/2003 Role of Pioglitazone in the Treatment of Nonalcoholic Steatohepatitis

1. PURPOSE/SPECIFIC AIMS To determine the role of pioglitazone in the treatment of nonalcoholic steatohepatitis (NASH) in patients with glucose intolerance or type 2 diabetes mellitus (T2DM). NASH is a disease characterized by elevated plasma aminotransferases and histopathological changes in liver characterized by hepatocellular steatosis, chronic inflammation and fibrosis (1-3). Pioglitazone, a new thiazolidinedione (TZD), has proven to be safe and effective for the treatment of type 2 diabetes mellitus (T2DM) (4). NASH affects ~10-20% of obese and type 2 diabetic subjects (1-3, 5, 6). While the pathogenesis of NASH is poorly understood, there is consensus that insulin resistance and its associated abnormalities in lipid metabolism play a key role in the development of liver fat accumulation, and TNF-alpha is a major mediator in the progression of liver damage (7-9). Currently, there is no satisfactory therapy for NASH.

Pioglitazone improves insulin sensitivity and glycemic control in patients with T2DM (4, 10-12), but the mechanism of action of TZDs is unclear (13, 14). Pioglitazone activates genes involved in lipid synthesis, causing a reduction in plasma free fatty acid (FFA) and triglycerides (15). TZDs decrease excessive triglyceride accumulation in liver (16), muscle (17), and visceral fat (11, 16, 18), with a redistribution of fat to subcutaneous adipose stores (14). TZDs also antagonize the metabolic effects of TNF-alpha (19-22). Because pioglitazone ameliorates insulin resistance, reverses the metabolic abnormalities that contribute to hepatic fat infiltration (increased plasma glucose, FFA, and triglyceride concentrations), and antagonizes the effects of TNF-alpha, it follows that pioglitazone may prove useful for the treatment of patients with NASH.

In order to evaluate this hypothesis, we plan to treat for 6 months a group of patients with impaired glucose tolerance (IGT) or T2DM with pioglitazone in a randomized, double-blinded, placebo-controlled trial. Three major endpoints will be measured before and after treatment (see Methods for a detailed description):

1. Liver histologic response; assessed by liver biopsy. Steatosis and inflammatory changes will be quantified using a standardized staging system.
2. Liver fat content: measured by liver magnetic resonance spectroscopy (MRS).
3. Hepatic insulin sensitivity and glucose metabolism: Because fat infiltration of liver and muscle causes insulin resistance and impairs glucose tolerance, we will measure parameters of metabolic control including fasting plasma glucose, free fatty acids, fructosamine, HbA1c and fasting lipid profile. To assess the effect of pioglitazone on hepatic insulin sensitivity, fasting (basal) and postprandial hepatic glucose production will be studied using a double-tracer technique (infusion of 3-3H glucose combined with an oral glucose load radiolabeled with 1-14C glucose) (23). Glucose and lipid oxidation will be measured by indirect calorimetry (24). In addition, an index of hepatic and peripheral insulin sensitivity will be derived from the oral glucose tolerance test (OGTT) (25).

ELIGIBILITY:
Inclusion Criteria:

1. Be able to communicate meaningfully with the Investigator and be legally competent to provide written informed consent.
2. Patients must have an age range between 21 to 70 years (inclusive).
3. NASH confirmed by liver biopsy.
4. Subjects must meet the criteria for impaired glucose tolerance (FPG concentration <126 mg/dl and a two hour plasma glucose value during the oral glucose tolerance test [OGTT] ≥140 but <200 mg/dl) or type 2 diabetes mellitus (FPG concentration ≥ 126 mg/dl or a two hour plasma glucose value during the OGTT ≥200 mg/dl) (62). Subjects with a FPG greater than 260 mg/dl will be excluded from the study.
5. Diabetic patients will be allowed to be on sulfonylureas or repaglinide but not on metformin, a thiazolidinedione or insulin. Patients must have been on a stable dose of allowed chronic medications for four weeks prior to entering the double-blind treatment period.
6. Female patients must be non-lactating and must either be at least two years post-menopausal, or be using adequate mechanical contraceptive precautions (i.e. intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period. Patients on oral contraceptives or an hormonal implant will be excluded.
7. All participants must have the following laboratory values:

Hemoglobin ≥ 13 gm/dl in males, or

≥ 12 gm/dl in females WBC count ≥ 3,000/mm3 Neutrophil count ≥ 1,500/mm3 Platelets ≥ 100,000/mm3 Prothrombin time within 3 seconds of control Albumin ≥3.0 g/dl Serum creatinine ≤ 1.6 mg/dl Creatinine phosphokinase ≤ 2 times upper limit of normal AST (SGOT) ≤ 2.5 times upper limit of normal ALT (SGPT) ≤ 2.5 times upper limit of normal Alkaline phosphatase ≤ 2.5 times upper limit of normal

Exclusion Criteria:

1. Any cause of chronic liver disease other than NASH (such as -but not restricted to- alcohol or drug abuse, medication, chronic hepatitis B or C, autoimmune, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency).
2. Any clinical evidence or history of ascitis, bleeding varices, or spontaneous encephalopathy.
3. No past (for at least for 1 year) or current history of alcohol abuse (alcohol consumption greater than one drink per day).
4. Prior surgical procedures to include gastroplasty, jejuno-ileal or jejunocolic bypass.
5. Prior exposure to organic solvents such as carbon tetrachloride.
6. Total parenteral nutrition (TPN) within the past 6 months.
7. Diabetics with a FPG greater than 260 mg/dl on initial visit.
8. Diabetics who are taking metformin, a thiazolidinedione or insulin.
9. Subjects with type 1 diabetes mellitus.
10. Patients on chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for 4 weeks before entry into the study. Patients on estrogens or other hormonal replacement therapy, tamoxifen, raloxifene, oral glucocorticoids or chloroquine will be excluded.
11. Patients with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation), will not be studied.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-10; Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Liver histology (Kleiner criteria, Hepatology 2005) | 6 months.

SECONDARY OUTCOMES:
Liver fat content by MRS. | 6 months.
Double-tracer OGTT (EGP, glucose clearance). | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cusi, MD, Principal Investigator — University of Texas
Locations (1):
- Audie L Murphy VA Hospital, San Antonio, Texas, United States

REFERENCES:
- [Background] Cusi K. Thiazolidinediones in NASH. An odd couple meant to be? J Clin Gastroenterol. 2009 Jul;43(6):503-5. doi: 10.1097/MCG.0b013e3181a15e51. No abstract available. PMID 19384246
- [Result] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Result] Balas B, Belfort R, Harrison SA, Darland C, Finch J, Schenker S, Gastaldelli A, Cusi K. Pioglitazone treatment increases whole body fat but not total body water in patients with non-alcoholic steatohepatitis. J Hepatol. 2007 Oct;47(4):565-70. doi: 10.1016/j.jhep.2007.04.013. Epub 2007 May 24. PMID 17560678
- [Result] Gastaldelli A, Harrison SA, Belfort-Aguilar R, Hardies LJ, Balas B, Schenker S, Cusi K. Importance of changes in adipose tissue insulin resistance to histological response during thiazolidinedione treatment of patients with nonalcoholic steatohepatitis. Hepatology. 2009 Oct;50(4):1087-93. doi: 10.1002/hep.23116. PMID 19670459
- [Result] Ali R, Cusi K. New diagnostic and treatment approaches in non-alcoholic fatty liver disease (NAFLD). Ann Med. 2009;41(4):265-78. doi: 10.1080/07853890802552437. PMID 19353360
- [Result] Cusi K. Nonalcoholic fatty liver disease in type 2 diabetes mellitus. Curr Opin Endocrinol Diabetes Obes. 2009 Apr;16(2):141-9. doi: 10.1097/MED.0b013e3283293015. PMID 19262374